CLINICAL TRIAL: NCT03497702
Title: Phase II Study of Neo-adjuvant Chemotherapy With Letrozole in Patients With Estrogen Receptor Positive/HER-2 Negative Breast Cancer
Brief Title: Neo-adjuvant Chemotherapy With Letrozole in Patients With Estrogen Receptor Positive/HER-2 Negative Breast Cancer
Acronym: NeoChAI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Keun Seok Lee, Head, Center for Breast Cancer, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2017-0110
Record Dates: First submitted 2018-03-18; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer; Invasive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Docetaxel; Letrozole; Leuprolide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Patients receive neoadjuvant chemotherapy (doxorubicin 60mg/m2 IV and cyclophosphamide 600mg/m2 IV on day 1 every 3 weeks for 4 cycles followed by docetaxel 75mg/m2 IV on day 1 every 3 weeks for 4 cycles) plus letrozole with or without leuproelin depending on menopausal status
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Letrozole; Drug: leuprorelin

INTERVENTIONS:
Drug: Doxorubicin — 60mg/m2 IV every 3 weeks for 4 cycles
Drug: Cyclophosphamide — 600mg/m2 IV every 3 weeks for 4 cycles
Drug: Docetaxel — 75mg/m2 IV every 3 weeks for 4 cycles
Drug: Letrozole — 2.5 mg once daily preoperably
Drug: leuprorelin — 3.75 mg SC every 4 weeks for premenopausal patients

SUMMARY:
This is an exploratory interventional study that initiates chemotherapy with letrozole in patients with estrogen receptor positive/HER2-negative breast cancer preoperably.

DETAILED DESCRIPTION:
STUDY RATIONALE: Patients with ER+/HER2- operable breast cancers who are candiate of neoadjuant chemotherapy generally receive chemotherapy alone before operation, followed by adjuvant endocrine therapy. Because endocrine therapy is primarily delivered in the postoperative setting, the ability to add the efficacy of aromatase inhibitors combined with chemotherapy is lost. This study offers the unique opportunity to assess the synergistic or additive responsiveness of breast tumors to endocrine therapy plus chemotherapy while the tumors are still in vivo by treating patients with an aromatast inhibitor combined with chemotherapy before surgery and assessing pCR rates.

PRIMARY OBJECTIVE: The primary objective is to determine the frequency of pCR in breast and axilla.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven breast cancer patients who are candidate of neoadjuvant chemotherapy with AC followed by Docetaxel
* Age: 19-70 years
* ER or PR positive ,cT2-3N0 or cT1-3/N+ M0 (ER-positive ≥1% nuclear staining by immunohistochemistry , Allred score≥3 )
* Available FFPE tissue for biomarker study
* HER2-negative by ASCO/CAP guideline
* Patients who agree to adequate contraception
* ECOG scores of 0-2
* Normal or acceptable kidney, liver, cardiovascular, and bone marrow functions
* Patients who provide consent

Exclusion Criteria:

* Inflammatory breast cancer
* Distant metastasis
* Cerebral vascular accidents including transient ischemic attack
* Pulmanary thromboembolism or deep vein thrombosis with 6 months; however, patients who received more than 6 weeks of anticoagulation within 6 months and remains asymptomatic are eligible.
* With a history of malignant tumor or complicated with other malignant tumors in addition to breast cancer, except for non-melanoma skin cancer, curatively resected early gastric cancer, differentiated thyoid cancer < 1 cm, or other cured malignant tumor without recurrence for at least 3 years
* Ejection Fraction <55% by MUGA scan / Echo CG
* No available tissue for biomarker study
* Pregnant or lactating women
* Patients with other serious diseases or medical conditions: Pituitary adenoma, Malabsorption syndrome, Major resection of gastrointestinal tract, Corrected QT interval > 480 msec, Congestive heart failure or unstable angina pectoris, myocardial infarction, stent insertion, angioplasty, coronary bypass surgery, symptomatic peripheral artery disease within 6 months before the enrollment
* NYHA class III or IV congestive heart failure
* Uncontrolled hypertension and uncontrolled high-risk arrhythmia considered by the investigator
* Major surgery, major trauma, and/or unhealed wound, fracture, or ulcer within 4 weeks
* Acute hemorrhage or hemorrhagic tendency
* Obvious neurological or psychiatric disorders, including psychosis, epileptic dementia and other diseases which may affect the understanding and sign of the informed consent
* Uncontrolled acute infection
* Patients with allergic constitution and any known or suspected drug allergy
* Concurrent use of other investigational drugs; or participating in other clinical trials involving investigational drugs within 30 days before this study
* Patients with mental illness or other conditions affecting the patient compliance
* Not suitable for the trial considered by the investigator

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete remission (pCR) | within 6 weeks following the last dose of chemotherapy
  pCR defined as no invasive residuals in breast and lymph nodes (ypT0/Tis, ypN0 [MD Anderson definition])

SECONDARY OUTCOMES:
Adverse events | during 6 months of neoadjuvant chemotherapy
  Frequency and severity of hematological and non-hematological adverse events and laboratory abnormalities according to Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Response rate | during 6 months of neoadjuvant chemotherapy
  Overall objective clinical response rate = CR + PR rate, measured by MRI (or US) and assessed by RECIST criteria.
Downstaging to breast conserving surgery (BCS) | within 6 weeks following the last dose of chemotherapy
  Ratio of the number of patients with breast conserving surgery converted from planned mastectomy over the number of patients with initially planned mastectomy
Disease free survival | Patients will be followed up to 6 years
  Disease-free survival (DFS) following operation.

CONTACTS AND LOCATIONS:
Overall Officials: Keun Seok Lee, MD, PhD, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided